CLINICAL TRIAL: NCT03409809
Title: Implementation Support for Prevention Program Delivery by College Peer Educators
Acronym: PI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Stanford University (Other); University of Texas at Austin (Other); Trinity University, Texas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MH112743
Record Dates: First submitted 2017-12-07; First posted 2018-01-24 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Eating Disorder
Keywords: Implementation Support; Eating Disorder; Dissemination; Prevention; Peer Leader
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training Alone (Experimental): This condition involves an intensive 2-day initial train-the-trainer workshop that simultaneously trains peer educators to deliver the intervention and campus supervisors to train and support future peer educators, plus the facilitator guide and facilitator support website.
  Interventions: Behavioral: Training
- Training and Technical Assistance (Experimental): This condition involves an intensive 2-day initial train-the-trainer workshop that simultaneously trains peer educators to deliver the intervention and campus supervisors to train and support future peer educators, plus the facilitator guide and facilitator support website. This condition additionally contains a 1/2 day implementation training to articulate goals, needs, leadership structure, adoption options, recruitment strategies, and communication.
  Interventions: Behavioral: Training and Technical Assistance
- Training, Tech. Assist., Qual. Assurance (Experimental): This condition involves an intensive 2-day initial train-the-trainer workshop that simultaneously trains peer educators to deliver the intervention and campus supervisors to train and support future peer educators, plus the facilitator guide and facilitator support website. This condition additionally contains a 1/2 day implementation training to articulate goals, needs, leadership structure, adoption options, recruitment strategies and communication. Furthermore, this condition will have 1 year of technical assistance, coaching, and quality assurance to enhance implementation skills and sustainability.
  Interventions: Behavioral: Training, Tech. Assistance, Quality Assurance/Improvement

INTERVENTIONS:
Behavioral: Training — Level of Support: Intensive 2-day train-the-trainer workshop, facilitator guide and facilitator support website.
  Arms: Training Alone
Behavioral: Training and Technical Assistance — Level of Support: Intensive 2-day train-the-trainer workshop, facilitator guide, and facilitator support website, plus half-day implementation training to further define goals, needs, leadership structure and strategy for adoption and recruitment.
  Arms: Training and Technical Assistance
Behavioral: Training, Tech. Assistance, Quality Assurance/Improvement — Level of Support: As for "Training and Technical Assistance" arm, plus 1-year of technical assistance, coaching, and quality assurance to enhance skills for implementation and sustainability.
  Arms: Training, Tech. Assist., Qual. Assurance

SUMMARY:
This project will evaluate 3 approaches of implementation support for university peer leaders who will deliver a prevention program with a particularly strong evidence-base compared to changes observed in outcomes in response to usual care at the universities before implementation. This study aims to advance knowledge of this innovative and economical way to provide college prevention programs to reduce the burden of mental illness in the college student population.

DETAILED DESCRIPTION:
Several interventions for mental health problems are efficacious and effective, but few are routinely offered to college students, who represent 59% of young adults. This is regrettable because college students are at high risk for mental health problems (e.g., depression, substance abuse, eating disorders), and college counseling centers lack sufficient clinicians to offer individual therapy to all afflicted students and are not well positioned to deliver prevention programs. One solution for this service shortfall is to have peer educators deliver scripted group-based prevention programs, which can more efficiently reduce the burden of mental illness than individual therapy. Targeting college students is a cost-effective tactic for delivering prevention programs and has vast potential reach because 85% of colleges have peer educator programs. Peer educators have effectively delivered several prevention programs, sometimes producing larger effects than clinicians. This study will investigate 3 levels of implementation support (training, training with technical assistance, and training with technical assistance and quality assurance) and the impacts of differing levels of implementation support on program outcomes across 57 college campuses nationwide. Specifically we have five aims for this study:

Aim 1: Test whether greater implementation support is associated with graded increases in fidelity and competence in delivering the scripted prevention program. This will be assessed by an established procedure for reliably rating fidelity and competence of audio-recorded intervention sessions.

Aim 2: Test whether greater implementation support, which should increase fidelity and competence of intervention delivery, is associated with graded increases in student attendance of intervention sessions (recorded by the peer educators) and effectiveness of the prevention program (measured by pre-to-post changes in core outcomes assessed with anonymous surveys completed by group participants) and compared to parallel pre-to-post change data collected from students at the colleges before implementation is initiated.

Aim 3: Test whether greater implementation support is associated with graded increases in program reach (% of female students at each college who complete the prevention program during the 1-year implementation period) and sustainability (% of female students at each college who complete the prevention program during the subsequent 2-year sustainability monitoring period).

Aim 4: Test whether Consolidated Framework for Implementation of Research (CFIR) indices of perceived intervention factors, outer and inner setting factors, peer educator attributes, and process factors after the initial training correlate with fidelity, competence, attendance, effectiveness, and reach over the 1-year implementation period and with sustainability. We will test whether at the end of the initial implementation period the 3 conditions differ on relevant CFIR indices and on the progress and speed of implementation.

Aim 5: Compare the prevention program delivery cost in the 3 implementation conditions, and the relative cost-effectiveness of each condition in terms of attaining fidelity, competence, attendance, and effectiveness, reach, and sustainability, plus cost-savings from and reductions in waitlists and eating disorder prevalence at clinics.

Starting in March of 2020, virtually-hosted Body Project groups are being recommended to participating Peer Education teams in contexts where in-person groups can not be offered due to COVID-19 social distancing guidelines. Existing research indicates that virtual Body Project groups are a viable and effective alternative in-person groups.

ELIGIBILITY:
Five Categories of Study Participant: (1) Peer Educator, (2) Peer Educator Supervisor, (3) Clinician, (4) Body Project Group Participant, (5) Usual Care Participant

1. Peer Educator

   Inclusion Criteria:
   * College undergraduate student Peer Educators with an interest in promoting body satisfaction
   * Willing to attend a 2-day Body Project train-the-trainer (TTT) training

   Exclusion Criteria:
   * Undergraduate college students from a college or university* that does not have a formal Peer Education Program
2. Peer Educator Supervisor

   Inclusion Criteria:
   * College or University* staff members with an interest in promoting body satisfaction
   * Willing to attend a 2-day Body Project train-the-trainer (TTT) training

   Exclusion Criteria:
   * Not a staff member
3. Clinician

   Inclusion Criteria:
   * Clinician working at a US College or University*

   Exclusion Criteria:
   * Not a clinician
4. Body Project Group Participant

   Inclusion Criteria:
   * College* students with an interest in promoting body satisfaction

   Exclusion Criteria:
   * Not a college student
5. Usual Care Participant

Inclusion Criteria:

* College* students with an interest in promoting body satisfaction

Exclusion Criteria:

* Not a College* student
* Current or past participant in a Body Project group

  * Participating students and staff are randomized at the school level.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2261 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Fidelity of Program Implementation as assessed by 25-item Session Adherence Scale (Stice et al., 2013a) | 12 months
  Peer educators' adherence to scripted intervention manual and accuracy of script delivery as coded through evaluation of audio-recorded sessions by two clinicians independently coding a random selection of sessions using the Session Adherence Scale. Coders will indicate the extent to which peer leaders adhere to the 25 total total necessary components of the 4-session intervention script using a scoring guide ranging from 10 (indicating no adherence) to 100 (indicating perfect adherence) with a possible total score range of 250 to 2500. Inter-rater agreement for Session Adherence Scale has been found to be .92 (Stice et al., 2013a).
Competence of Program Implementation as assessed by 12-item Group Leader Competence Scale (Stice et al., 2013a) | 12 months
  Peer educators' competence with intervention delivery as assessed by 12-item Group Leader Competence Scale measuring various indicators of a competent group facilitator (e.g. leaders allot equal speaking time for all members.) Coders will indicate the extent to which peer leaders show competence in their delivery of the scripted intervention across 12 items using a scoring guide ranging from 10 (indicating poor competence) to 100 (indicating superior competence) with a possible total score range of 120 to 1200. Inter-rater agreement for Group Leader Competence Scale has been found to be .96 (Stice et al., 2013a).

SECONDARY OUTCOMES:
Attendance | 12 months
  Attendance levels of participants as recorded by peer educators
Reach | 12 months
  Percentage of students who complete the prevention program at 1 year post-educator training
Sustainability | 24 months
  Percentage of students who complete the prevention program during the subsequent 2-year sustainability monitoring period
Delivery Cost | 12 months
  Dollar amount delivery cost for each arm of the implementation support model
Relative Cost-Effectiveness | 12 months, 24 months
  Relative cost-effectiveness of each arm of the implementation support model
Perceived Characteristics of the Intervention as measured by the 28-item Provider Intervention Adoption Scale | 1 Week or less post training
  Perceived Characteristics of the Intervention as measured by the 28-item Provider Intervention Adoption Scale. Respondents will indicate their level of agreements with the 27 items using a 5-point Likert-type scale ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree) with a possible score ranging from 27 to 135.
Project Knowledge | Baseline, 1 week or less post-training, 12 months
  Peer educators' declarative project knowledge as measured by the 20-item Body Project Knowledge Scale. Peer educators will indicate whether the statements in this scale are "true" or "false," with a possible score ranging from 0 for no correct replies to 20 for every answer correct.
Provider Attitudes Towards Evidence-Based Interventions | Baseline, 1 week or less post-training, 12 months
  Provider Attitudes Towards Evidence-Based Interventions as measured by the 50-item Evidence-Based Practice Attitude Scale (EBPAS-50), which will assess provider attitudes toward adopting evidence-based intervention (Aarons, 2004); it has four subscales: Appeal (intuitive appeal of evidence-based interventions), Requirements (likelihood of adopting evidence-based interventions given supervisor, organizational, or system requirements), Openness (general openness to new practices), and Divergence (perceived divergence between research developed interventions and current practice), which sum up to a total score representing respondents' global attitude toward adopting and using evidence-based practice. Respondents will indicate the extent to which they agree with each item on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very great extent). A higher total score indicates a more positive attitude toward adopting and using evidence-based practice. 23 items are reverse-scored.
Implementation Progress | Baseline, 12 months
  Implementation Progress as measured by the Prevention Implementation Progress Scale
Peer Educator Self-Efficacy | Baseline, 1 week or less post-training, 12 months
  Peer Educator Self-Efficacy as measured by the 14-item Peer Educator Self-Efficacy Questionnaire. Respondents will degree of confidence on a 6-point scale ranging from 1 (No Confidence) to 6 (Complete Confidence). Scores will range from 14 (no demonstrated peer educator self-efficacy) to 84 (high peer educator self-efficacy.)
Inner Setting | Baseline, 12 months
  Inner Setting sub domains assessed using the Team Climate Inventory
Outer Setting | Baseline
  Evaluate presence or absence of formal policies related to evidence-based programs, fiscal and other organizational resources for peer educators based on two coded interviews

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Oregon Research Institute, Eugene, Oregon
  - University of Texas at Austin, Austin, Texas
  - Trinity University, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duru C, Bearman SK, Rohde P, Shaw H, Stice E. A qualitative study of modifications and adaptations to an evidence-based prevention intervention during implementation on college campuses. Eat Disord. 2025 Apr 30:1-17. doi: 10.1080/10640266.2025.2497638. Online ahead of print. PMID 40305559
- [Derived] Bearman SK, Rohde P, Pauling S, Gau JM, Shaw H, Stice E. Predictors of the sustainability for an evidence-based eating disorder prevention program delivered by college peer educators. Implement Sci. 2024 Jul 4;19(1):47. doi: 10.1186/s13012-024-01373-9. PMID 38965587
- [Derived] Stice E, Rohde P, Gau JM, Shaw H. Implementation factors that predict larger effects from a peer educator delivered eating disorder prevention program at universities. J Consult Clin Psychol. 2023 Feb;91(2):60-70. doi: 10.1037/ccp0000783. Epub 2023 Feb 23. PMID 36821334